CLINICAL TRIAL: NCT05130775
Title: Measurement of Tricuspid Regurgitation Volume for Assessment of Tricuspid Regurgitation Using 3D Transesophageal Echocardiography
Status: Withdrawn | Type: Observational
Why Stopped: The study was stopped due to non availability of sample for data collection
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00001677
Record Dates: First submitted 2021-11-15; First posted 2021-11-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transesophageal echocardiograpgy — 3D acquisition of the right ventricle regurgitation volume

SUMMARY:
This study is a prospective observational chart review. The aim of the study is to evaluate tricuspid regurgitation volume using 3D volumetric assessment as an accurate method for tricuspid regurgitation severity in comparison to VCA.

ELIGIBILITY:
Inclusion Criteria:

-All degrees of tricuspid regurgitation minimal, mild, moderate and severe will be included

Exclusion Criteria:

* Exclusion criteria will be non-sinus rhythm, more than mild pulmonary regurgitation, more than trace aortic regurgitation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18 years and older with all grades of tricuspid regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Tricuspid regurgitation volume | 12 months
  We will evaluate patients with different grades TR by both 3DVCA and the 3D volumetric approach

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes